CLINICAL TRIAL: NCT02279966
Title: An Interventional, Randomised, Double-blind, Parallel-group, Placebo-controlled, Active-referenced (Paroxetine), Fixed-dose Study on the Efficacy of Vortioxetine on Cognitive Dysfunction in Working Patients With Major Depressive Disorder
Brief Title: Efficacy of Vortioxetine on Cognitive Dysfunction in Working Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15906A; 2014-000230-34 (EudraCT Number)
Record Dates: First submitted 2014-10-21; First posted 2014-10-31 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine; Paroxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vortioxetine 10 mg (Experimental): daily, encapsulated, orally
  Interventions: Drug: Vortioxetine 10 mg
- Paroxetine 20 mg (active reference) (Other): daily, encapsulated, orally
  Interventions: Drug: Paroxetine 20 mg
- Placebo (Placebo Comparator): capsules, orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vortioxetine 10 mg
  Other Names: Brintellix®; Lu AA21004
  Arms: Vortioxetine 10 mg
Drug: Paroxetine 20 mg
  Arms: Paroxetine 20 mg (active reference)
Drug: Placebo
  Arms: Placebo

SUMMARY:
To assess the efficacy of acute treatment with 10 mg/day vortioxetine versus placebo on cognitive performance (focusing on the aspect concerning speed of processing, executive functioning, attention) in working patients with major depressive disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* The patient has MDD, diagnosed according to Diagnostic and Statistical Manual of Mental Disorders, 4th edition, Text Revision (DSM-IV-TR™) recurrent major depressive disorder (MDD) (classification 296.3x).
* The patient has a MADRS total score ≥26.
* The patient has had the current major depressive episode (MDE) for ≥3 months.
* The patient is aged ≥18 and ≤65 years.
* The patient is employed full or part-time (defined as minimum 50% full time working hours per week). Part time work should not be due to a medical or mental illness other than MDD.
* The patient has been in the current job/position for at least 3 months.
* The patient has no plans to change jobs or retire within treatment period.
* The patient is not on a sick leave, and at the Screening and Randomisation Visits, there are no plans to send the patient on a sick leave.
* The patient is not receiving disability benefits.

Exclusion criteria:

* The patient has a score ≥70 on the DSST (number of correct symbols) at the Baseline Visit.
* The patient is, in the opinion of the investigator, not able to complete the neuropsychological tests validly at the Baseline Visit.
* The patient has physical, cognitive, or language impairment of such severity as to adversely affect the validity of the data derived from the neuropsychological tests.
* The patient is diagnosed with reading disability (dyslexia).
* The patient has a history of lack of response to previous adequate treatment with vortioxetine or paroxetine.
* The patient has any current psychiatric disorder or Axis I disorder (according to DSM-IV-TR™ criteria) other than MDD, as assessed using MINI.
* The patient has a current or has had a diagnosis of dysthymic disorder within 3 months preceding the onset of current episode (DSM-IV-TR™ criteria).
* The patient has borderline, schizotypal, schizoid, paranoid, or histrionic, antisocial personality disorders (axis II) as comorbid or primary diagnosis (DSM-IV-TR™ criteria).
* The patient suffers from personality disorders, mental retardation, pervasive development disorder, attention-deficit/hyperactivity disorder, organic mental disorders, or mental disorders due to a general medical condition (DSM-IV-TR™ criteria).
* The patient has a current diagnosis or history of manic or hypomanic episode, schizophrenia or any other psychotic disorder, including major depression with psychotic features (DSM-IV-TR™ criteria).

Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in Digit Symbol Substitution Test (DSST): number of correct symbols | Baseline to Week 8

SECONDARY OUTCOMES:
Change in Trail Making Test (TMT) score: TMT-A; speed of processing | Baseline to Week 8
Change in TMT-B; executive functioning | Baseline to Week 8
Change in reaction time score: Choice Reaction Time (CRT); attention | Baseline to Week 8
Change in reaction time score: Simple Reaction Time (SRT); psychomotor speed) | Baseline to Week 8
Change in Stroop Colour Naming Test (STROOP): incongruent score; executive functioning | Baseline to Week 8
Change in STROOP: congruent score; speed of processing | Baseline to Week 8
Change in Perceived Deficits Questionnaire - Depression (PDQ-D) total score | Baseline to Week 8
Change in Montgomery and Asberg Depression Rating Scale (MADRS) total score | Baseline to Week 8
Change in Clinical Global Impression - Severity of Illness (CGI-S) | Baseline to Week 8
Clinical Global Impression - Global Improvement (CGI-I) score | Week 8
Change in the Functioning Assessment Short Test (FAST) total score | Baseline to Week 8
Change in University of San Diego Performance-based Skills Assessment - Brief (UPSA-B) total score | Baseline to Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (18):
- Estonia (3):
  - EE001, Tallinn
  - EE002, Tallinn
  - EE004, Võru
- Finland (5):
  - FI002, Helsinki
  - FI003, Helsinki
  - FI001, Kuopio
  - FI008, Oulu
  - FI007, Tampere
- Germany (5):
  - DE002, Berlin
  - DE001, Bielefeld
  - DE003, Frankfurt
  - DE007, Frankfurt
  - DE008, Schwerin
- Lithuania (5):
  - LT002, Kaunas
  - LT006, Palanga
  - LT003, Šilutė
  - LT001, Vilnius
  - LT005, Vilnius

REFERENCES:
- [Derived] Christensen MC, Sluth LB, McIntyre RS. Validation of the University of California San Diego Performance-based Skills Assessment (UPSA) in major depressive disorder: Replication and extension of initial findings. J Affect Disord. 2019 Feb 15;245:508-516. doi: 10.1016/j.jad.2018.11.034. Epub 2018 Nov 5. PMID 30439678
- See also: EMA EudraCT Results: 2014-000230-34 — https://www.clinicaltrialsregister.eu/ctr-search/trial/2014-000230-34/results